CLINICAL TRIAL: NCT03437317
Title: Emotional Perceptual Training as a Treatment for Social Anxiety: Behavioral and Neural Evidence.
Acronym: PTL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Wen Li, Dr. Wen Li, Associate Professor of Psychology and Neuroscience, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTL-2017.21521
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Anxiety Disorders and Symptoms; Social Anxiety Disorder
Keywords: Social Anxiety; Threat processing; Magnetoencephalography (MEG)
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either an active training group or a control group. The active participants completed 8 blocks of a perceptual training task, while the control group performed 8 blocks of a gender discrimination task
  that received the perceptual retraining protocol
Who Masked: Participant
Masking Description: Participants were blind to their assigned condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Active - MEG (Experimental): Participants completed 1 session of 8 Perceptual Retraining blocks following an instructional presentation.
  Interventions: Behavioral: Perceptual Retraining
- Control - MEG (Sham Comparator): Participants completed 1 session of 8 blocks of Gender Discrimination Task.
  Interventions: Behavioral: Gender Discrimination
- Active - 3 Behavior/EEG (Experimental): Participants completed 3 sessions of Perceptual Retraining following an instructional presentation. The first session included 6 blocks of perceptual training, and the second session included 12 blocks of perceptual training. No perceptual training was performed in session 3. Sessions were spaced approximately 7 days apart, with a minimum of 3 days and a maximum of 14 days apart.
  Interventions: Behavioral: Perceptual Retraining
- Active - 1 Behavior/MEG (Experimental): Participants completed 1 session of 6 Perceptual Retraining blocks following an instructional presentation.
  Interventions: Behavioral: Perceptual Retraining
- Control - 3 Behavior/MEG (Sham Comparator): Participants completed 3 sessions of a Gender Discrimination Task. The first session included 6 blocks of gender discrimination task, and the second session included 12 blocks of the gender discrimination task. No gender discrimination task was performed in session 3. Sessions were spaced approximately 7 days apart, with a minimum of 3 days and a maximum of 14 days apart.
  Interventions: Behavioral: Gender Discrimination

INTERVENTIONS:
Behavioral: Perceptual Retraining — Participants viewed faces varying in their expression of anger and were asked to identify if the face was angry or neutral via button press. Participants were provided with feedback if their categorization of the face as neutral or angry was correct. Each participant was assigned 4 levels of angry faces based on their decision point of anger detection in faces. Faces were selected based on the closest existing anger morph to the category boundary; for example, a decision point of 40% anger was closest to the 38% anger face, and so the faces used would have been 17%, 31%, 45%, and 59% anger. For this example, responses of "neutral" to the 31% angry face would be marked as correct, whereas a similar response to the 45% angry face would be incorrect, as it was above their decision point.
  Arms: Active - 1 Behavior/MEG; Active - 3 Behavior/EEG; Active - MEG
Behavioral: Gender Discrimination — Participants viewed faces varying in their expression of anger and were asked to identify if the face was male or female via button press.
  Arms: Control - 3 Behavior/MEG; Control - MEG

SUMMARY:
The Perceptual Training Study is a series of studies performed with the purpose of identifying a potential avenue for treatment of mood disorders, particularly anxiety-based mood disorders. The underlying theme is that neural representations may be threat-oriented, and may also be generalized to non-threatening cues by means of similarity to threatening representations. These may result in anxiety symptoms from innocuous cues. The idea behind the perceptual training is to create a divorce between the threat representations and cues which should be considered non-threatening, enhancing perceptual acuity and potentially reducing anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Normal or corrected-to-normal vision

Exclusion Criteria:

* History of a diagnosed neurological or Diagnostic and Statistical Manual of Mental Disorders - IV Axis I disorder
* Currently taking prescribed psychoactive drugs, including anti-depressants or anxiolytics.
* Having electrically, magnetically, or mechanically activated implants (e.g. cardiac pacemakers), due to incompatibility with MRI and MEG systems.
* Pregnancy or suspected pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Behavioral Evidence for Categorical Perception Changes | Baseline to Study Completion (14 to 28 Days)
  Participants will be asked to respond if they detected anger in faces varying in their levels of anger expression. This task is used to determine a perceptual bias for threat/anger in faces that is related to increases in social anxiety symptoms, and assess for improvements in the categorization of angry vs. neutral faces. that align with modulations of neural responses (MEG and EEG evidence) indexing perceptual processing of the faces following perceptual retraining.
Neural Evidence for Categorical Perception Changes | Baseline to Study Completion (14 to 28 Days)
  Neural activity will be recorded using EEG and MEG to measure neural processes underpinning categorical perception of anger in faces. Changes in this neural perceptual index will be assessed following perceptual retraining to provide a neural mechanism underpinning behavioral improvements in perceptual categorization and subsequent reductions in anxiety.

SECONDARY OUTCOMES:
Social Anxiety Symptoms - Social Phobia Scale | Baseline to Study Completion (14 to 28 Days)
  Change in social anxiety symptomatology through perceptual retraining
Social Anxiety Symptoms - Liebowitz Social Anxiety Scale | Baseline to Study Completion (14 to 28 Days)
  Change in social anxiety symptomatology through perceptual retraining

IPD SHARING:
Plan to Share IPD: Undecided